CLINICAL TRIAL: NCT03720795
Title: Parent-Led Stepped-Care Cognitive-Behavioral Treatment for Youth With ASD and Co-occurring Anxiety
Brief Title: Stepped-Care Cognitive-Behavioral Treatment for Youth With ASD and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Eric A Storch, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCM SC-CBT001
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Cognitive Behavioral Therapy; Autism Spectrum Disorder; Anxiety Disorders; Obsessive-Compulsive Disorder; Social Anxiety Disorder; Generalized Anxiety Disorder; Specific Phobia
MeSH Terms: conditions — Autism Spectrum Disorder; Anxiety Disorders; Obsessive-Compulsive Disorder; Phobia, Social; Generalized Anxiety Disorder; Phobia, Specific

STUDY DESIGN:
Intervention Model Description: Single group observational.
Masking Description: The rater is unaware of treatment status, that is if the child continues to receive treatment after Step 1 (versus being in maintenance).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stepped Care CBT (Other): Stepped Care CBT consists of two main steps. Step One involves 4 parent-led, therapist-assisted treatment sessions, up to 45 minutes each, over an 8-week period. Participants who do not show significant improvement in symptom severity at the end of Step One, are then 'stepped up' to receive Step Two, which involves 12 weekly, therapist-led, parent-assisted treatment sessions, up to 60 minutes each.
  Interventions: Behavioral: Stepped Care CBT

INTERVENTIONS:
Behavioral: Stepped Care CBT — Stepped Care CBT is a multi-method, parent-led approach, consisting of two main steps. Step one involves a "low-intensity" delivery of CBT, consisting of more flexible, parent-led, at-home treatment. Participants who do not show improvement in symptom severity at the end of Step One, are then "stepped up" to receive Step Two. Step two involves a "high intensity" delivery of CBT, consisting of therapist-led, parent-assisted weekly treatment sessions.

SUMMARY:
This study implements a parent-led, flexible, individually-tailored cognitive-behavioral intervention for children with ASD and anxiety.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) affects as many as 1 out of 59 individuals, with many higher-functioning youth not diagnosed until school-age or later. This equates to ~102,000 children under the age of 14 years in the state of Texas alone. Significant impairment in social and adaptive functioning are common, as are comorbid behavioral health disorders, with anxiety disorders affecting between 50-80% of youth with ASD. Given the relative frequency of anxiety disorders among children with ASD, the associated impairment, and worsening trajectory over time without intervention, there is a great need for treatment that specifically addresses anxiety-related symptoms in ASD. Cognitive-behavioral therapy (CBT) has been established as a first-line treatment for anxiety disorders among youth with and without ASD. A particular form of CBT, Behavioral Intervention for Anxiety in Children with ASD (BIACA), has demonstrated efficacy in a number of studies. However, treatment is delivered by therapists as "full-packages" (i.e., 12-16 clinic sessions), which can be therapist-intensive, costly, impractical for families, and not responsive to parental preferences. Alternatives approaches, such as parent-led, stepped-care models that improve accessibility, are efficient, provide personalized care, and lower mental health treatment cost, are greatly needed. Stepped-care models provide a lower-intensity first step (e.g., parent-led, less costly, and more convenient for parents) as the initial treatment with the assumption that a proportion of individuals will respond to the first step and others will need to step up to more intensive treatment. Matching treatment to families' needs and tailoring subsequent treatment may be an efficient and effective approach, as well as consistent with parents' desire to help their child. Given this, together with the substantial impairment associated with clinical anxiety in individuals with ASD across the age span, this study implements a parent-led, flexible, individually-tailored cognitive-behavioral intervention for children with ASD and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Child is between the ages 4-14 years at consent/assent.
* The child meets criteria for ASD.
* The child meets criteria for clinically significant anxiety and/or OCD symptoms.
* Anxiety and/or OCD is the primary presenting problem.
* One parent/guardian is able and willing to attend.
* The child has a Full Scale and Verbal Comprehension Intelligence Quotient >70.

Exclusion Criteria:

* The child has a diagnosis of lifetime DSM-5 bipolar disorder, psychotic disorder, and/or intellectual disability.
* The child has severe current suicidal/homicidal ideation and/or self-injury requiring medical intervention.
* The child is receiving concurrent psychotherapy for anxiety.
* Initiation of a psychotropic medication less than 4 weeks prior to study enrollment or a stimulant/psychoactive medication less than 2 weeks prior to study enrollment.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were not pre-assigned to groups. If participants did not respond to Step One of treatment, then they were stepped up to Step Two. Those who did respond to treatment at Step One then they entered a maintenance phase
Period: Phase 1
Arm/Group | Stepped Care CBT
Started | 76
Completed | 64
Not Completed | 12
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 6
Not completed — Protocol Violation | 1
Not completed — Other | 1
Period: Phase 2
Arm/Group | Stepped Care CBT
Started | 64
Entered Maintenance | 20
Stepped Up to Step 2 | 44
Completed | 47
Not Completed | 17
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 10
Not completed — Protocol Violation | 2
Period: 3 Month Follow Up
Arm/Group | Stepped Care CBT
Started | 47
Entered Maintenance | 18
Stepped Up to Step 2 | 27
Completed | 45
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Of the 76 participants, 64 entered phase two of the study. Of these 64, 20 entered the maintenance phase (were responders to Step One) and 44 stepped up to Step Two
Groups:
- Stepped-Care CBT: Stepped Care CBT consists of two main steps. Step One involves 4 parent-led, therapist-assisted treatment sessions, up to 45 minutes each, over an 8-week period. Participants who do not show significant improvement in symptom severity at the end of Step One, are then 'stepped up' to receive Step Two, which involves 12 weekly, therapist-led, parent-assisted treatment sessions, up to 60 minutes each.
  Stepped Care CBT: Stepped Care CBT is a multi-method, parent-led approach, consisting of two main steps. Step one involves a "low-intensity" delivery of CBT, consisting of more flexible, parent-led, at-home treatment. Participants who do not show improvement in symptom severity at the end of Step One, are then "stepped up" to receive Step Two. Step two involves a "high intensity" delivery of CBT, consisting of therapist-led, parent-assisted weekly treatment sessions.
Arm/Group | Stepped-Care CBT
Number analyzed (Participants) | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 76
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.86 (2.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26
  Not Hispanic or Latino | 50
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 57
  More than one race | 6
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 76
Clinical Global Impressions - Severity [Mean (Standard Deviation); unit: units on a scale] — Clinician-rated child psychopathology severity rating. A single item is scored 0-6 (0= no illness; 6= extremely severe symptoms).
  units on a scale | 3.66 (1.07)
Pediatric Anxiety Rating Scale (PARS) [Mean (Standard Deviation); unit: units on a scale] — Clinician-rated child anxiety severity throughout the past week. Each item is scored on a 0 to 5 scale (higher scores correspond to greater severity), yielding a total between 0 and 35.
  units on a scale | 21.54 (3.91)

OUTCOME MEASURES:

1. Primary Outcome: 7-item Pediatric Anxiety Rating Scale
Description: Clinician rated child anxiety severity throughout the past week. Each item is scored on a 0 to 5 scale (higher scores correspond to greater severity), yielding a total between 0 and 35.
Time Frame: Baseline (before treatment), mid-treatment (on average 12 weeks), post-treatment (on average 24 week), 3 month follow up; Post-treatment scores are reported.
Population: 48 participants completed either the maintenance phase or Step Two of treatment
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stepped Care CBT
Number analyzed (Participants) | 48
Score on a scale | 11.87 (6.93)

2. Primary Outcome: Clinical Global Impression-Improvement
Description: Clinician rated child psychopathology improvement since initial rating. A single item is scored 0-6 (0 = very much worse; 6= very much improved).
Time Frame: Mid-treatment (on average 12 weeks), post-treatment (on average 24 week), 3 month follow up; Post-treatment scores are reported.
Population: 48 participants were considered completers of Step 2 or the Maintenance Phase. The count is the number of participants that are considered "much improved" or "very much improved" on the CGI-I
Measure: Count of Participants; unit: Participants
Arm/Group | Stepped Care CBT
Number analyzed (Participants) | 48
Participants | 42

3. Secondary Outcome: Clinical Global Impression-Severity
Description: Clinician rated child psychopathology severity rating. A single item is scored 0-6 (0= no illness; 6= extremely severe symptoms).
Time Frame: as for outcome 1
Population: 48 participants either completed Step Two or the maintenance phase.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stepped Care CBT
Number analyzed (Participants) | 48
Score on a scale | 1.88 (.98)

ADVERSE EVENTS:
Time Frame: Participants were enrolled in the study for up to 9 months, which is the same time as when adverse event data were collected
Description: The definition of an adverse event is the same as found on clinicaltrials.gov
Groups:
- Stepped Care CBT: Stepped Care CBT consists of two main steps. Step One involves 4 parent-led, therapist-assisted treatment sessions, up to 45 minutes each, over an 8-week period. Participants who do not show significant improvement in symptom severity at the end of Step One, are then 'stepped up' to receive Step Two, which involves 12 weekly, therapist-led, parent-assisted treatment sessions, up to 60 minutes each.
  Stepped Care CBT: Stepped Care CBT is a multi-method, parent-led approach, consisting of two main steps. Step one involves a "low-intensity" delivery of CBT, consisting of more flexible, parent-led, at-home treatment. Participants who do not show improvement in symptom severity at the end of Step One, are then "stepped up" to receive Step Two. Step two involves a "high intensity" delivery of CBT, consisting of therapist-led, parent-assisted weekly treatment sessions.
  All Adverse Event reports are combined here as there is only one group that is split into two milestones of "Entered Maintenance" or "Stepped Up to Step 2"
Arm/Group | Stepped Care CBT
All-Cause Mortality (participants affected / at risk) | 0/76
Serious Adverse Events (participants affected / at risk) | 0/76
Other Adverse Events (participants affected / at risk) | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-04-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT03720795/Prot_SAP_ICF_000.pdf